CLINICAL TRIAL: NCT06369740
Title: Case and Use Scenario Study to Gain Knowledge on the User Needs for a Medical Device for Hemophilia a Monitoring
Status: Completed | Type: Observational
Sponsor: Enzyre B.V. (Industry)
Collaborators: Indiana Hemophilia & Thrombosis Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: ENZ20-2024-INDIANAPOLIS
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Hemophilia a
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Hemophilia A patients - case scenario focus groups: 60 patients with hemophilia A aged 12 years and older that partake in the case scenario focus groups
  Interventions: Other: Case scenarios - questionnaire; Other: Case scenarios - Focus groups
- Healthcare providers - case scenario focus groups: 30 healthcare providers with experience in the field of hemophilia A that partake in the case scenario focus groups
  Interventions: Other: Case scenarios - questionnaire; Other: Case scenarios - Focus groups
- Hemophilia A patients - use scenarios: 6 patients with hemophilia A aged 12 years and older that partake in the use scenarios usability evaluation
  Interventions: Other: Use scenarios - Usability test; Other: Use scenarios - interview
- Healthcare providers - use scenarios: 6 healthcare providers with experience in the field of hemophilia A that partake in the use scenarios usability evaluation
  Interventions: Other: Use scenarios - Usability test; Other: Use scenarios - interview

INTERVENTIONS:
Other: Case scenarios - questionnaire — Participants fill in a questionnaire on the current care of hemophilia A and envisioned use scenarios of a point-of-care diagnostic device for hemophilia A.
  Groups: Healthcare providers - case scenario focus groups; Hemophilia A patients - case scenario focus groups
Other: Case scenarios - Focus groups — Participants partake in focus groups on the current care for hemophilia A, the envisioned use scenarios of point-of-care diagnostic device for hemophilia A and desired features of such a diagnostic device.
  Groups: Healthcare providers - case scenario focus groups; Hemophilia A patients - case scenario focus groups
Other: Use scenarios - Usability test — Participants are asked to perform basic tasks with the mock-ups with minimal instructions, they will also be given a graphic of the user interface (GUI).
  Groups: Healthcare providers - use scenarios; Hemophilia A patients - use scenarios
Other: Use scenarios - interview — The participants will be interviewed and asked for their opinions and experiences with the mock-ups.
  Groups: Healthcare providers - use scenarios; Hemophilia A patients - use scenarios

SUMMARY:
This observational study consists of two parts.

In part one, case scenario focus groups with hemophilia A patients and healthcare providers (HCPs) will be held. This parts aims to identify potential use scenarios of a point of care (POC) in vitro medical for patients with hemophilia A. The main questions it aims to answer are:

* How is coagulation lab testing for patients with hemophilia A currently organized?
* What is the interest and what are desired alternatives of a POC in-vitro diagnostic medical device for patients with hemophilia A?

Part two of the study consists of a use scenario study in which patients with hemophilia A and HCPs will evaluate two types of non-functional mock-ups of a POC in vitro medical device. The main goal of this part is to evaluate the usability of the current prototypes of the POC device.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* With Hemophilia A diagnosis
* All Hemophilia A severity categories are eligible (mild, moderate, or severe)
* Aged 12 years and older
* For children aged 12 through 17 their parent must provide permission by signing the informed consent form
* Consider English their primary language (capable of communicating in English verbally and in writing)
* Capable of giving informed consent or assent

Family member(s) of patients:

* Related to a patient with Hemophilia A (mild, moderate, or severe)
* Aged 18 years and older
* Consider English their primary language (capable of communicating in English verbally and in writing)
* Capable of giving informed consent or assent

Healthcare professionals:

* Healthcare workers specialized in hemophilia care. (e.g. hematologists, nurse practitioners, physician assistants, nurses, and pharmacists)
* Capable of giving informed consent

Exclusion Criteria:

Patients:

* Without a diagnosis of Hemophilia A
* With acquired Hemophilia A
* Younger than 12 years of age
* Unable to communicate in English
* Incapable of giving consent or assent for themselves

Specifically for the case scenario focus group

* Unwilling to consent to voice recording
* Participating in the use scenario part of the study

Specifically for the use scenario part of the study

* Unwilling to consent to video recording
* Participating in the case scenario part of the study

Family members:

* No relation to a patient with Hemophilia A (mild, moderate, or severe)
* Related to a patient with acquired Hemophilia A
* Younger than 18 years of age
* Unable to communicate in English
* Incapable of giving consent or assent for themselves

Specifically for the case scenario focus group

* Unwilling to consent to voice recording
* Participating in the use scenario part of the study

Specifically for the use scenario part of the study

* Unwilling to consent to video recording
* Participating in the case scenario part of the study

Healthcare professionals:

* Without any prior hematological experience
* Not licensed as hematologists, nurse practitioners, physician assistants, nurses or pharmacists
* Unable to communicate in English
* Incapable of giving their consent to participate

Specifically for the case scenario part of the study • Unwilling to consent to voice recording

Specifically for the use scenario part of the study

• Unwilling to consent to video recording

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients or caregivers of patients with hemophilia A of any severity (mild, moderate, severe) aged 12 years and older are considered. Patients have tbe able to speak English and have give informed consent. In patients ages 12-17, parents will also have to give informed consent. Patients are not allowed to participate in both the use scenarios and the case scenarios parts of the study.
  Healthcare providers specialized in hemophilia care are also included. This could be hematologists, nurse practitioners, physician assistents, nurses and pharmacists.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2024-08-22 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Current management of Hemophilia A coagulation lab testing | One day
  Themes regarding the current management of Hemophilia A coagulation lab testing
Potential case scenarios for a point of care in-vitro diagnostic device for hemophilia A | One day
Usability issues of the current POC in-vitro diagnostic device prototypes | one day
  Overview of identified usability issues

SECONDARY OUTCOMES:
User preferences for the point of care in-vitro diagnostic device | One day
Problems with current Hemophilia A coagulation monitoring | One day
Potential benefits of a POC device for home use, near-patient use or in clinic use | One day

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana Hemophilia & Thrombosis Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No